CLINICAL TRIAL: NCT04365387
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Assess Immunization Responses in Adult and Adolescent Subjects With Moderate-to-Severe Atopic Dermatitis Treated With Nemolizumab
Brief Title: A Study to Assess Immunization Responses in Adult and Adolescent Participants With Moderate-to-Severe Atopic Dermatitis Treated With Nemolizumab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RD.06.SPR.118380
Record Dates: First submitted 2020-04-24; First posted 2020-04-28 (Actual); Results first posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Dermatitis, Atopic
Keywords: Eczema; AD; Vaccine; Nemolizumab; Pruritis; Itchy
MeSH Terms: conditions — Dermatitis, Atopic; Eczema; Pruritus | interventions — nemolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nemolizumab (Experimental): Participants received a loading dose of nemolizumab (60 milligram [mg]) via 2 subcutaneous (SC) injections at baseline. Nemolizumab (30 mg) was administered via a single subcutaneous injection every 4 weeks (Q4W) at Weeks 4, 8, and 12.
  Interventions: Drug: Nemolizumab
- Placebo (Placebo Comparator): Participants received a placebo via 2 SC injections at baseline. Placebo was administered via a single subcutaneous injection Q4W at Weeks 4, 8, and 12.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nemolizumab — Nemolizumab was administered by 2 SC injections as 60-mg loading dose at baseline and a single 30-mg dose at Weeks 4, 8, and 12.
  Arms: Nemolizumab
Drug: Placebo — Placebo was administered by 2 SC injections at baseline and a single dose at Weeks 4, 8, and 12.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the effect of nemolizumab (CD14152) on humoral immune responses to tetanus and meningococcal vaccination in adult and adolescent participants with moderate-to-severe atopic dermatitis (AD).

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, multi-center, parallel-group study in adult and adolescent participants (≥ 12 to 54 years) with moderate-to-severe AD. Eligible participants must have a documented history of inadequate response to topical AD medication(s). Approximately 200 participants were randomized 1:1 to receive either 30 mg nemolizumab (with a 60 mg loading dose) or placebo, stratified by baseline disease severity Investigator Global Assessment (IGA) (IGA = 3, moderate; IGA = 4, severe). The study consisted of a 2- to 4-week screening period, a 16-week treatment period, and an 8-week follow-up period (12 weeks after the last study drug injection).

ELIGIBILITY:
Inclusion Criteria:

* Chronic AD for at least 2 years
* EASI score >= 16
* IGA score >= 3
* AD involvement >= 10% of BSA
* Peak (maximum) pruritus NRS score of at least 4.0

Exclusion Criteria:

* Body weight < 30 kilogram (kg)
* History of hypersensitivity (including anaphylaxis) to an immunoglobulin product (plasma-derived or recombinant, eg, monoclonal antibody) or to any of the study drug excipients
* History of severe allergic reaction to either vaccine or to vaccine components including alum, thimerosal, phenol
* Participants for whom administration of the meningococcal vaccine provided in this study is contraindicated or medically inadvisable
* Participants for whom administration of the tetanus, diphtheria, and pertussis vaccine provided in this study is contraindicated or medically inadvisable
* Receipt of any vaccine (except inactivated influenza vaccine) within 12 weeks prior to screening, any meningococcal vaccine within 1 year prior to screening, or any tetanus-, diphtheria-, or pertussis-containing vaccine within 5 years prior to screening

Ages: 12 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 242 (Actual)
Dates: Start 2020-03-05 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-07-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (63):
- United States (63):
  - Galderma Investigational Site (Site#9922), Phoenix, Arizona
  - Galderma Investigational Site (Site#8873), Scottsdale, Arizona
  - Galderma Investigational Site (Site#8447), Fort Smith, Arkansas
  - Galderma Investigational Site (Site#8831), Anaheim, California
  - Galderma Investigational Site (Site#8854), Canoga Park, California
  - Galderma Investigational Site (Site#8578), Cerritos, California
  - Galderma Investigational Site (Site#8791), Fresno, California
  - Galderma Investigational Site (Site#8845), Huntington Beach, California
  - Galderma Investigational Site (Site#8833), Inglewood, California
  - Galderma Investigational Site 2 (Site#8833), Inglewood, California
  - Galderma Investigational Site (Site#8858), Long Beach, California
  - Galderma Investigational Site (Site#8130), Los Angeles, California
  - Galderma Investigational Site (Site#8813), Los Angeles, California
  - Galderma Investigational Site (Site#8837), Pomona, California
  - Galderma Investigational Site (SIte#8870), Boca Raton, Florida
  - Galderma Investigational Site (Site#8786), Clearwater, Florida
  - Galderma Investigational Site (Site#8792), Doral, Florida
  - Galderma Investigational Site (Site#8391), Hialeah, Florida
  - Galderma Investigational Site (Site#8836), Jacksonville, Florida
  - Galderma Investigational Site (Site#8850), Margate, Florida
  - Galderma Investigational Site (Site#8851), Miami, Florida
  - Galderma Investigational Site (Site#9921), Miami Lakes, Florida
  - Galderma Investigational Site (Site#8840), Ocoee, Florida
  - Galderma Investigational Site (Site#8788), Orlando, Florida
  - Galderma Investigational Site (Site#8213), Ormond Beach, Florida
  - Galderma Investigational Site (Site#8856), Ormond Beach, Florida
  - Galderma Investigational Site (Site#8843), Sweetwater, Florida
  - Galderma Investigational Site (Site#8764), Tampa, Florida
  - Galderma Investigational Site 2 (Site#8816), Tampa, Florida
  - Galderma Investigational Site (Site#8839), Tampa, Florida
  - Galderma Investigational Site (Site#8739), Normal, Illinois
  - Galderma Investigational Site (Site#8142), Indianapolis, Indiana
  - Galderma Investigational Site (Site#8532), Overland Park, Kansas
  - Galderma Investigational Site (Site#8812), Metairie, Louisiana
  - Galderma Investigational Site (Site#8793), Towson, Maryland
  - Galderma Investigational Site (Site#8033), Clinton Township, Michigan
  - Galderma Investigational Site (Site#8129), Fort Gratiot, Michigan
  - Galderma Investigational Site (Site#8849), Troy, Michigan
  - Galderma Investigational Site (Site#8876), Bridgeton, Missouri
  - Galderma Investigational Site (Site#8847), Las Vegas, Nevada
  - Galderma Investigational Site (Site#8848), Las Vegas, Nevada
  - Galderma Investigational Site 2 (Site#8864), Las Vegas, Nevada
  - Galderma Investigational Site (Site#8420), Portsmouth, New Hampshire
  - Galderma Investigational Site (Site#9924), Raritan, New Jersey
  - Galderma Investigational Site (Site#8828), Kew Gardens, New York
  - Galderma Investigational Site (Site#9919), Raleigh, North Carolina
  - Galderma Investigational Site (Site#8795), Shelby, North Carolina
  - Galderma Investigational Site (Site#8857), Oklahoma City, Oklahoma
  - Galderma Investigational Site (Site#8841), Medford, Oregon
  - Galderma Investigational Site (Site#8428), Philadelphia, Pennsylvania
  - Galderma Investigational Site (Site#8353), Yardley, Pennsylvania
  - Galderma Investigational Site (Site#8777), Charleston, South Carolina
  - Galderma Investigational Site (Site#8200), Goodlettsville, Tennessee
  - Galderma Investigational Site (Site#8846), Austin, Texas
  - Galderma Investigational Site (Site#8855), Beaumont, Texas
  - Galderma Investigational Site (Site#8245), Dallas, Texas
  - Galderma Investigational Site (Site#8868), Houston, Texas
  - Galderma Investigational Site (Site#8817), Katy, Texas
  - Galderma Investigational Site (Site#8787), Plano, Texas
  - Galderma Investigational Site (Site#8329), San Antonio, Texas
  - Galderma Investigational Site (Site#8003), Webster, Texas
  - Galderma Investigational Site (Site#8844), Orem, Utah
  - Galderma Investigational Site (Site#9935), Springville, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 42 sites in United states from 05 Mar 2020 to 07 Jul 2023.
Pre-assignment Details: A total of 242 participants were randomized and out of which only 234 received treatment in the study.
Groups:
- Nemolizumab: Participants received a loading dose of nemolizumab (60 milligram [mg]) via 2 subcutaneous (SC) injections at baseline. Nemolizumab (30 mg) administered via a single subcutaneous injection every 4 weeks (Q4W) at Weeks 4, 8, and 12. Participants also received single doses of Tdap and MCV4 vaccines at week 12.
- Placebo: Participants received a placebo (matching to Nemolizumab) via 2 SC injections at baseline. Placebo was administered via a single subcutaneous injection Q4W at Weeks 4, 8, and 12. Participants also received single doses of Tdap and MCV4 vaccines at week 12.
Period: Overall Study
Arm/Group | Nemolizumab | Placebo
Started | 123 | 119
Modified Intent to Treat (mITT) Population (Modified Intent-to-Treat (mITT) population consisted of all randomized participants who received at least one dose of study drug and vaccine injection, had an evaluable vaccine response and did not receive any systemic rescue therapy prior to the post-vaccination vaccine response assessment.) | 80 | 78
Safety Population (The Safety population consisted of all randomized subjects who received at least one administration of study drug. The treatment group assignment in this population was defined by the treatment actually received. This population was used for all the analyses of safety endpoints.) | 119 | 115
Completed | 90 | 93
Not Completed | 33 | 26
Not completed — Adverse Event | 4 | 2
Not completed — Participants request | 14 | 14
Not completed — Lost to Follow-up | 8 | 5
Not completed — Protocol deviation | 3 | 4
Not completed — Participant compliance with visit schedule | 1 | 0
Not completed — Participant incarcerated | 1 | 0
Not completed — Participant moved out of town (relocated) | 0 | 1
Not completed — Participant PEF not eligible per sponsor | 1 | 0
Not completed — Due to working hours, could not return to other visits | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat Population (ITT) population consisted of all randomized participants.
Groups:
- Nemolizumab: Participants received a loading dose of nemolizumab (60 mg) via 2 SC injections at baseline. Nemolizumab (30 mg) administered via a single SC injection Q4W at Weeks 4, 8, and 12. Participants also received single doses of Tdap and MCV4 vaccines.
- Placebo: Participants received a placebo (matching to Nemolizumab) via 2 SC injections at baseline. Placebo was administered via a single subcutaneous injection Q4W at Weeks 4, 8, and 12. Participants also received single doses of Tdap and MCV4 vaccines.
- Total: Total of all reporting groups
Arm/Group | Nemolizumab | Placebo | Total
Number analyzed (Participants) | 123 | 119 | 242
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.2 (11.62) | 32.1 (12.00) | 33.6 (11.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 69 | 147
  Male | 45 | 50 | 95
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 43 | 45 | 88
  Not Hispanic or Latino | 79 | 73 | 152
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 13 | 19 | 32
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 35 | 31 | 66
  White | 70 | 62 | 132
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Positive Serum Immunoglobulin G (IgG) Response (>= 4-Fold Increase or >= 0.2 IU/mL in Anti-Tetanus IgG Concentrations) to Tetanus Toxoid at Week 16 (4 Weeks Post-vaccination)
Description: Percentage of participants with a positive serum IgG response to tetanus toxoid, defined as greater than or equal to (>=) 4-fold increase in anti-tetanus IgG concentrations from baseline in participants with pre-vaccination anti-tetanus IgG concentrations >= 0.1 international unit per milliliter (IU/mL); or >= 0.2 IU/mL anti-tetanus IgG concentrations in participants with pre-vaccination antitetanus IgG concentrations less than (<) 0.1 IU/mL, at Week 16 (4 weeks post-vaccination) were reported.
Time Frame: At Week 16 (4 weeks post-vaccination)
Population: mITT population consisted of all randomized participants who received at least one dose of study drug and vaccine injection, had an evaluable vaccine response and did not receive any systemic rescue therapy prior to the post-vaccination vaccine response assessment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Nemolizumab | Placebo
Number analyzed (Participants) | 80 | 78
Percentage of Participants | 67.5 | 65.4
Statistical Analysis 1: Comparison: Nemolizumab vs Placebo; Test type: Other; Cochran-Mantel-Haenszel = 2.1, 90% CI 2-sided [-10.3 to 14.5] — Risk Difference (90% CI) were estimated using weighted average of stratum-specific proportion using Cochran-Mantel-Haenszel (CMH)

2. Secondary Outcome: Percentage of Participants With a Positive Serum IgG Response (>=2-Fold Increase or >= 0.2 IU/mL in Anti-tetanus IgG Concentrations) to Tetanus Toxoid at Week 16 (4 Weeks Post-vaccination)
Description: Percentage of participants with a positive serum IgG response to tetanus toxoid, defined as >= 2-fold increase in anti-tetanus IgG concentrations from baseline in participants with pre-vaccination anti-tetanus IgG concentrations >= 0.1 IU/mL; or >= 0.2 IU/mL anti-tetanus IgG concentrations in participants with pre-vaccination Anti tetanus IgG concentrations < 0.1 IU/mL, at Week 16 (4 weeks post-vaccination) were reported.
Time Frame: At Week 16 (4 weeks post-vaccination)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Nemolizumab | Placebo
Number analyzed (Participants) | 80 | 78
Percentage of Participants | 78.8 | 83.3
Statistical Analysis 1: Comparison: Nemolizumab vs Placebo; Test type: Other; Cochran-Mantel-Haenszel = -4.6, 90% CI 2-sided [-14.9 to 5.7] — Risk Difference (90% CI) were estimated using weighted average of stratum-specific proportion using CMH

3. Secondary Outcome: Percentage of Participants With Serum Anti-tetanus IgG Concentrations of >= 0.1 IU/mL at Week 16
Description: Percentage of participants with serum anti-tetanus IgG concentrations of >= 0.1 IU/mL at Week 16 were reported. The detection and characterization of antibodies to tetanus toxoid was performed using a validated immunoassay.
Time Frame: At Week 16
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Nemolizumab | Placebo
Number analyzed (Participants) | 80 | 78
Percentage of Participants | 100 | 100

4. Secondary Outcome: Percentage of Participants With Serum Anti-tetanus IgG Concentrations of >= 1.0 IU/mL at Week 16
Description: Percentage of participants with serum anti-tetanus IgG concentrations of >= 1.0 IU/mL at Week 16 were reported. The detection and characterization of antibodies to tetanus toxoid was performed using a validated immunoassay.
Time Frame: At Week 16
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Nemolizumab | Placebo
Number analyzed (Participants) | 80 | 78
Percentage of Participants | 97.5 | 96.2
Statistical Analysis 1: Comparison: Nemolizumab vs Placebo; Test type: Other; Cochran-Mantel-Haenszel = 1.4, 90% CI 2-sided [-3.2 to 5.9] — Risk Difference (90% CI) were estimated using weighted average of stratum-specific proportion using CMH

5. Secondary Outcome: Percentage of Participants With a Positive Serum Bactericidal Antibody (SBA) Response to Meningococcal Serogroup C (MenC) Polysaccharide at Week 16
Description: Percentage of participants with a positive SBA response to meningococcal serogroup C polysaccharide, defined as >= 4-fold increase in SBA reciprocal titer from baseline (using non-imputed values), at Week 16 (4 weeks postvaccination) were reported.
Time Frame: At Week 16
Population: mITT population consisted of all randomized participants who received at least one dose of study drug and vaccine injection, had an evaluable vaccine response and did not receive any systemic rescue therapy prior to the post-vaccination vaccine response assessment. Here "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Number; unit: Percentage of Participants
Arm/Group | Nemolizumab | Placebo
Number analyzed (Participants) | 61 | 66
Percentage of Participants | 77.0 | 63.6
Statistical Analysis 1: Comparison: Nemolizumab vs Placebo; Test type: Other; Cochran-Mantel-Haenszel = 13.3, 90% CI 2-sided [0.1 to 26.4] — Risk Difference (90% CI) were estimated using weighted average of stratum-specific proportion using CMH for non-Imputed values

6. Secondary Outcome: Percentage of Participants With a Positive SBA Response (Defined as SBA Reciprocal Titer ≥8) to MenC Polysaccharide at Week 16
Description: Percentage of participants with a positive SBA response to MenC polysaccharide, defined as SBA reciprocal titer >= 8, at Week 16 were reported. Immune response to meningococcal vaccination was determined by measuring functional antibody responses using an SBA assay.
Time Frame: At Week 16
Population: as for outcome 5
Measure: Number; unit: Percentage of Participants
Arm/Group | Nemolizumab | Placebo
Number analyzed (Participants) | 66 | 72
Percentage of Participants | 83.3 | 81.9
Statistical Analysis 1: Comparison: Nemolizumab vs Placebo; Test type: Other; Cochran-Mantel-Haenszel = 1.3, 90% CI 2-sided [-9.3 to 11.9] — Risk Difference (90% CI) were estimated using weighted average of stratum-specific proportion using CMH

ADVERSE EVENTS:
Time Frame: From Day 1 up to end of study (Week 24)
Description: Safety Population included all randomized participants who received at least one administration of study drug.
Groups:
- Placebo: Participants received a placebo via 2 SC injections at baseline. Placebo was administered via a single subcutaneous injection Q4W at Weeks 4, 8, and 12. Participants also received single doses of Tdap and MCV4 vaccines.
Arm/Group | Nemolizumab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/119 | 0/115
Serious Adverse Events (participants affected / at risk) | 0/119 | 1/115
Other Adverse Events (participants affected / at risk) | 44/119 | 38/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nemolizumab (N=119) | Placebo (N=115)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nemolizumab (N=119) | Placebo (N=115)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 13 | 6
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Superficial inflammatory dermatosis (Skin and subcutaneous tissue disorders) | 1 | 0
COVID-19 (Infections and infestations) | 4 | 2
Nasopharyngitis (Infections and infestations) | 1 | 1
Acute sinusitis (Infections and infestations) | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Root canal infection (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 1
Blood lactate dehydrogenase increased (Investigations) | 1 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0
Blood triglycerides increased (Investigations) | 0 | 1
Blood uric acid increased (Investigations) | 0 | 1
Electrocardiogram T wave amplitude decreased (Investigations) | 1 | 0
Lymphocyte count increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Peak expiratory flow rate decreased (Investigations) | 1 | 0
Urobilinogen urine increased (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Headache (Nervous system disorders) | 6 | 1
Somnolence (Nervous system disorders) | 1 | 1
Migraine (Nervous system disorders) | 1 | 0
Injection site pain (General disorders) | 1 | 1
Fatigue (General disorders) | 1 | 0
Injection site inflammation (General disorders) | 0 | 1
Injection site swelling (General disorders) | 1 | 0
Vaccination site pain (General disorders) | 0 | 1
Vessel puncture site bruise (General disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 3 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Eosinophilia (Blood and lymphatic system disorders) | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1
Penis injury (Injury, poisoning and procedural complications) | 0 | 1
Sunburn (Injury, poisoning and procedural complications) | 1 | 0
Proteinuria (Renal and urinary disorders) | 3 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Sweat gland tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Depression (Psychiatric disorders) | 1 | 1
Palpitations (Cardiac disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Vaccination site reaction (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-07-11): https://cdn.clinicaltrials.gov/large-docs/87/NCT04365387/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-15): https://cdn.clinicaltrials.gov/large-docs/87/NCT04365387/SAP_001.pdf